CLINICAL TRIAL: NCT00319189
Title: Efficacy and Safety of Nateglinide Treatment in Renal Treatment Recipients With Post Transplant Diabetes Mellitus or Impaired Glucose Tolerance
Brief Title: Efficacy and Safety of Nateglinide Treatment in Renal Transplant Recipients
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: University of Oslo School of Pharmacy (Other)
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: Starlix in RTR
Record Dates: First submitted 2006-04-27; First posted 2006-04-27 (Estimated); Last update posted 2006-05-10 (Estimated); Status verified 2006-04

CONDITIONS: Renal Transplant Recipients; Posttransplant Diabetes Mellitus; Posttransplant Impaired Glucose Tolerance
Keywords: Nateglinide; Renal; Kidney; Transplantation; Diabets; Glucose
MeSH Terms: interventions — Nateglinide

INTERVENTIONS:
Drug: Nateglinide

SUMMARY:
The objective of the present study is to evaluate both the efficacy and safet of nateglinide in renal transplanta recipients with posttransplant diabetes mellitus or impaired glucose tolerance. Primarily will the change in glucose tolerance and acute insuline responce be addressed.

ELIGIBILITY:
Inclusion Criteria:

* Reduced glucose tolerance (fasting glucose < 6.1 mmol/L AND 2 hour glucose between 6.7 and 9.9 mmol/L) or posttransplant diabetes mellitus (fasting glucose > 6.1 mmol/L OR 2 hour glucose between >= 10.0 mmol/L)
* Stable patients fgollowing renal transplantation, less than 25% variation in serum creatinine last week and serum creatinine < 200 micromol/L

Exclusion Criteria:

* Patients with indulin dependent diabetes mellitus before or after transplantation
* Planned change in daily prednisolone dose during the study period
* Haemoglobin < 8g/dL

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 15
Dates: Start 2002-11; Study Completion 2003-11

PRIMARY OUTCOMES:
Glucose tolerance
Insuline release

SECONDARY OUTCOMES:
Glucose oxidation
Postprandial hyperlipidemia
Glomerular filtration rate
HbA1C
Fasting glucose
Plasma nitric oxide
Plasma endothelin-1

CONTACTS AND LOCATIONS:
Overall Officials: Trond Jenssen, MD, PhD, Principal Investigator — Rikshospitalet, Section of Nephrology
Locations (1):
- Rikshospitalet, Section of Nephrology, Oslo, Norway